CLINICAL TRIAL: NCT02390180
Title: Sorting of Oral Sensations
Status: Completed | Type: Observational
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Richard Mattes, Distinguished Prof., Nutrition Sciences, Purdue University
Other Study IDs: 055040
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Taste Qualities; Primary Tastes

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sorting all tastes: This group will receive 15 samples to taste and sort into groups. The samples included: a blank solution, hexenoic acid, decenoic acid, oleic acid, linoleic acid, glucose, fructose, sodium chloride (2), citric acid, acetic acid, quinine, urea, monosodium glutamate, and inosine monophosphate.
  Interventions: Other: Tasting solutions
- Sorting bitter tastes: This group will receive 12 samples to taste and sort into groups. The samples included: blank solutions (2), decenoic acid, oleic acid, linoleic acid, quinine (2), urea (2),caffeine, sucrose octaacetate, and propylthiouracil.
  Interventions: Other: Tasting solutions

INTERVENTIONS:
Other: Tasting solutions — Participants will taste a variety of food grade compounds including: hexenoic acid, decenoic acid, oleic acid, linoleic acid, glucose, fructose, salt, citric acid, acetic acid, quinine, urea, caffeine, sucrose octaacetate, propylthiouracil, phenylthiocarbamide, monosodium glutamate, and inosine monophosphate.

SUMMARY:
Recent research indicates that fatty acids in food may have a taste. There is no lexicon to describe the sensation of the fatty acids, but participants frequently describe the sensation as bitter or sour. The proposed study will ask participants who have been screened for their ability to detect fatty acids to sort a variety of taste stimuli, including sweet, sour, salty, bitter, umami, and fatty acid tastes. Observing how the participants sort the stimuli will allow us to determine if the fatty acid taste is unique from other taste sensations.

DETAILED DESCRIPTION:
Panelists will be screened for their ability to discriminate 0.5% linoleic acid emulsion from the blank using two sequential tetrad tests. Panelists will wear nose clips during the tests. Panelists must successfully complete both tetrads in order to qualify for the study. Panelists who qualify for the full study will provide written informed consent as well as data on their ethnic background, age, and their habitual fat intake. Heights and weights will be measured.

After completing the screening tests and the demographic questions, panelists will receive 15 samples (for the first group: "All tastes sorting") or 12 samples (for the second group: "Bitters sorting"). When panelists receive the samples, they will be instructed to put on nose clips and keep the clips on for the duration of the test. Participants will be provided with water for rinsing their mouths as well as a cup to spit the samples into after tasting. Panelists will be provided with more water and additional spit cups as necessary. Next, panelists will be instructed to: "Taste each sample, spit it into the spit cup, and rinse with water. Then, sort the samples into groups you believe are similar. Groups may contain as many or as few samples as you desire. You may have as many or as few groups as you desire." Once they have decided on their groups, they will write in a description for each group and rate the group for its overall similarity. After finishing this initial sorting task, if panelists have more than two total groups, they will be instructed to select the two groups they believe are most similar to each other and combine them. If panelists still have more than two total groups, they will be instructed to combine the two most similar groups again. This will continue until panelists only have two groups remaining. At each level, panelists will rate the new, combined group for its overall similarity on a visual analog scale, as before.

Data from this sorting task will be compiled in to dissimilarity matrices for each participant, showing how many groups it took them before each sample was combined with each other sample. This data will be analyzed to determine if the fatty acid samples are similar or unique in sensation from other taste qualities.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (self report), normal taste function

Exclusion Criteria:

* Medication that alters taste sensation, failed to detect 0.5% linoleic acid emulsion, allergic to dairy or nuts

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy men and women at least 18 years of age, not on any medication that alters taste sensation, and not allergic to dairy or nut products (samples contained a dairy protein and some sugars that were processed in facilities that also process nuts). Participants also had to pass a screening test to determine they could detect 0.5% linoleic acid emulsion compared to a blank solution.
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Similarity of taste sensations | 1 visit (only visit)
  Participants sort the solutions into groups, and then combine the groups based on which samples are similar in oral sensation. This is used to determine how similar or different each sample is from the others. We are primarily interested in how the fatty acids (hexenoic acid, oleic acid, linoleic acid, and decenoic acid) are sorted, and whether they are distinct from other tastes.

SECONDARY OUTCOMES:
Effect of dietary fat on taste sensation sorting | 1 visit (only visit)
  Dietary records will be used to classify participants' diets as high or low in fat. The analysis of similarity among samples will be repeated and compared between these two groups. We are primarily interested in how the fatty acids (hexenoic acid, oleic acid, linoleic acid, and decenoic acid) are sorted, and whether they are distinct from other tastes.
Effect of genetic ability to taste propylthiouracil on taste sensation sorting | 1 visit (only visit)
  Participants will be classified by their ability to taste 6-n-propylthiouracil (using filter papers wil phenylthiocarbamide and using data from sorting the bitter compounds). Tasters and non-tasters of this compound will be compared in their sorting of the different solutions. This will be done for the Sorting Bitter tastes group only. We are primarily interested in how the fatty acids (hexenoic acid, oleic acid, linoleic acid, and decenoic acid) are sorted, and whether they are distinct from other tastes.
Effect of gender on taste sensation sorting | 1 visit (only visit)
  Sorting patterns by males and females will be compared as well. We are primarily interested in how the fatty acids (hexenoic acid, oleic acid, linoleic acid, and decenoic acid) are sorted, and whether they are distinct from other tastes.
Effect of BMI on taste sensation sorting | 1 visit (only visit)
  Sorting patterns by lean, overweight, and obese participants will be compared as well, using the data collected on height and weight to calculate body mass index. We are primarily interested in how the fatty acids (hexenoic acid, oleic acid, linoleic acid, and decenoic acid) are sorted, and whether they are distinct from other tastes.

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Mattes, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States